CLINICAL TRIAL: NCT00617331
Title: A Randomized, Double-Blind, Clinical Trial Evaluating the Immunogenicity of an Inactivated Influenza A/H9N2 Vaccine Among Healthy Adults With and Without Prior Exposure to Influenza A/H2N2
Brief Title: H9 Priming Study in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Robert Johnson, HHS/NIAID/DMID
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 06-0073; N01AI30039C; N01AI30039 (NIH)
Record Dates: First submitted 2008-02-14; First posted 2008-02-18 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Influenza
Keywords: vaccine, priming, influenza, flu, A/H9N2
MeSH Terms: conditions — Influenza, Human | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Dose 7.5 mcg (Experimental): 7.5 micrograms of vaccine administered on Day 0 and Day 28.
  Interventions: Biological: Subvirion inactivated influenza A/H9N2 (G9 variant) vaccine
- Dose 30 mcg (Experimental): 30 micrograms of vaccine administered on Day 0 and Day 28.
  Interventions: Biological: Subvirion inactivated influenza A/H9N2 (G9 variant) vaccine

INTERVENTIONS:
Biological: Subvirion inactivated influenza A/H9N2 (G9 variant) vaccine — Inactivated subvirion influenza A/chicken/Hong Kong/G9/97 (H9N2) vaccine administered via intramuscular (IM) injection, dose 7.5 or 30 micrograms.

SUMMARY:
The purpose of this research study is to determine whether prior exposure to A/H2N2 viruses is associated with better antibody (part of the immune system that fights infection) responses after vaccination with an A/H9N2 flu vaccine. The study will evaluate how much antibody is made to the influenza virus after H9N2 flu vaccination and how the body reacts to different strengths of the H9N2 flu vaccine. This information may guide vaccine development for this virus as well as other bird flu viruses that have infected humans. Study participants will include 120 healthy subjects, age 18-38 or 44-59 years. Two different dosages of vaccine will be given in the muscle of the upper arm about 1 month apart. The assignment of vaccines to participants is governed by chance. Study procedures may include medical history, physical exam, and blood samples. Study participation duration is about 7 months.

DETAILED DESCRIPTION:
Influenza A viruses have the potential to cause worldwide epidemics and/or pandemics resulting in significant morbidity and mortality. The goals of this study are to determine whether persons over 44 years of age (born before 1964) have evidence of priming to influenza A/H9N2 viruses as measured by responses to two different dosage levels of an A/H9N2 vaccine. Evidence of priming for persons born before 1964 has implications in pandemic preparedness planning in that such individuals may need only a single vaccination to induce immunity compared to persons who are not immunologically primed. This study will also explore the immunogenicity of two-dose regimen using a homologous A/H9N2 virus as an antigen for the hemagglutination inhibition assay (HAI) and neutralizing antibody assays. Approximately 120 healthy adults will be enrolled into this single-center, randomized, double-blind trial of subvirion inactivated influenza A/H9N2 (G9 variant) vaccine given by intramuscular (IM) injection. Subjects will be stratified by age, with 50 percent in each dosage group being between the ages of 18 and 38 inclusive and the other 50 percent being between the ages of 44 and 59 years, inclusive. Subjects will be randomized 1:1 to receive 2 doses one month apart of one of two dosages (7.5 micrograms or 30 micrograms) of A/chicken/Hong Kong/G9/97 subvirion vaccine. The subjects and staff responsible for assessing responses after vaccination will be blinded to the dosage level that is administered. All subjects will receive two doses of their assigned dosage level given by the IM route separated by approximately 28 days. Subjects will be observed in the clinic for approximately 20 minutes after vaccination. Subjects will maintain a memory aid recording oral temperature, and systemic and local adverse events for 7 days after each inoculation. They will return to clinic on day 8 after vaccination (window 8-10) for adverse event (AE) assessment, concomitant medication assessment, a targeted physical exam (if indicated), and review of memory aid. AE data will be captured Day 0 through Day 56. Serious adverse event (SAE) data will be captured from Day 0 through the end of the trial (7 months after the first dose of vaccine). Serum for immunogenicity evaluations will be obtained prior to the first vaccination, at Day 0, prior to the second vaccination, at Day 28 and at Day 56. The primary objective is to determine whether persons 44-59 years of age show evidence of immunologic priming to A/H9 virus compared to persons 18-38 years of age. The secondary objectives are to evaluate dose-related immunogenicity 4 weeks after each vaccination and to evaluate the safety and tolerability of the vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female (as indicated by a negative urine pregnancy test immediately prior to vaccine administration) between the ages of 18 and 38 years, inclusive, or 44-59 years, inclusive.
* Women of childbearing potential who are at risk of becoming pregnant must agree to practice adequate contraception (e.g., barrier method, abstinence, and licensed hormonal methods) from at least 30 days prior to enrollment and for at least 3 months after receipt of dose 2.
* Be in good health, as determined by vital signs (heart rate less than 100 beats per minute, blood pressure systolic less than or equal to 140 mm Hg and greater than or equal to 90 mm Hg; diastolic less than or equal to 90 mm Hg, oral temperature less than 100 degrees Fahrenheit), medical history and a targeted physical examination based on medical history. (Stable medical condition - no change in prescription medication, dose or frequency of medication in the last 3 months and health outcomes of the specific disease are considered to be within acceptable limits in the last 6 months. Any change that is due to change of health care provider, insurance company etc, or that is done for financial reasons, as long as in the same class of medication will not be considered a violation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome will not be considered a violation of this inclusion criterion.)
* Able to understand and comply with planned study procedures.
* Provide informed consent prior to initiation of any study procedures and be available for all study visits.

Exclusion Criteria:

* Has a known allergy to eggs or other components of the vaccine including thimerosal.
* Has a positive urine pregnancy test prior to vaccination (if female of childbearing potential), is breast-feeding, or has the intention to become pregnant within 3 months of receipt of their second dose of vaccine.
* Is undergoing immunosuppression as a result of an underlying illness or treatment.
* Has an active neoplastic disease or a history of any hematologic malignancy.
* Is using oral or parenteral steroids, high-dose inhaled steroids (greater than 800 micrograms/day of beclomethasone dipropionate or equivalent) or other immunosuppressive or cytotoxic drugs.
* Has a history of receiving immunoglobulin or other blood product within the 3 months prior to enrollment in this study.
* Has a diagnosis of schizophrenia, bipolar disease or other major psychiatric diagnosis.
* Has received any other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrollment in this study.
* Has an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of responses (this includes, but is not limited to: known chronic liver disease, significant renal disease, unstable or progressive neurological disorders, diabetes mellitus, and transplant recipients).
* Has a history of severe reactions following immunization with contemporary influenza virus vaccines.
* Has an acute illness, including an oral temperature greater than 100.4 degrees Fahrenheit, within 1 week of vaccination.
* Has received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to each vaccination in the study, or expects to receive an experimental agent during the 7-month study period.
* Prior receipt of influenza A/H9N2 vaccine, other than the present study.
* Is planning to enroll in another clinical trial at any time during the study period (approximately 7 months total).
* Has known active human immunodeficiency virus, hepatitis B or hepatitis C infection.
* Has a history of alcohol or drug abuse in the last 5 years.
* Has a history of Guillain-Barré syndrome.
* Have been hospitalized for psychiatric illness, history of suicide attempt or confinement for danger to self or others.
* Are receiving psychiatric drugs (aripiprazole, clozapine, ziprasidone, haloperidol, molindone, loxapine, thioridazine, thiothixene, pimozide, fluphenazine, risperidone, mesoridazine, quetiapine, trifluoperazine, trifluopromazine, chlorprothixene, chlorpromazine, perphenazine, olanzapine, carbamazepine, divalproex sodium, lithium carbonate or lithium citrate). Subjects who are receiving a single antidepressant drug and stable for at least 3 months prior to enrollment, without de-compensating symptoms will be allowed to be enrolled in the study.
* Plan to travel outside of the USA in the time between the first vaccination and 56 days following the first vaccination.
* Has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
* Has any condition that the investigator believes may interfere with successful completion of the study.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2008-02; Primary Completion 2008-08 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Frequency of 4-fold or greater serum hemagglutination inhibition assay (HAI) and neutralizing antibody rises in both age groups to the homologous vaccine antigen. | 28 Days after the first vaccine dose.

SECONDARY OUTCOMES:
Frequencies of 4-fold or greater increase in titer between pre- and post-immunization samples. | 28 days after the second vaccination (day 56).
Frequencies and severity of solicited and local and systemic adverse events in each vaccine dosage/age group. | 7 days after each inoculation.
Proportion of subjects in each age/vaccine dosage group that achieves an HAI titer of at least 32. | 28 days after each vaccination (Day 28, Day 56).
Frequencies and GMT of serum HAI and serum neutralizing antibody against a homologous A/H9N2 virus. | One month after each vaccination (Day 28, Day 56).
Adverse event (AE) or serious adverse event (SAE) information (solicited in-clinic and via memory aids and periodic targeted physical assessment). | Duration of study.
Proportion of subjects in each group with serum HAI or neutralizing antibody to influenza A/H2N2 viruses and the frequency and magnitude of antibody responses. | Before and after vaccination.
Geometric mean titer (GMT) of serum HAI and serum neutralizing antibody against the influenza A/H9N2 virus. | One month after each vaccination (Day 28, Day 56).

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States